CLINICAL TRIAL: NCT02539849
Title: Effect of Prebiotic Fructo-oligosaccharides (FOS) on Intestinal Abundance of Faecalibacterium Prausnitzii in Patients With Crohn´s Disease
Brief Title: Effect of Prebiotic FOS on Intestinal Abundance of Faecalibacterium Prausnitzii in Patients With Crohn´s Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADA-FOS
Record Dates: First submitted 2015-08-04; First posted 2015-09-03 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adalimumab + FOS (Other): Adalimumab will be administered during 12 weeks in combination with daily FOS 6g. (FOS administration will start 2 weeks before Adalimumab)
  Interventions: Dietary Supplement: FOS; Drug: Adalimumab

INTERVENTIONS:
Dietary Supplement: FOS
Drug: Adalimumab

SUMMARY:
FOS improve gut colonization by Faecalibacterium prausnitzii in patients with Crohn's disease

DETAILED DESCRIPTION:
To demonstrate that FOS increases counts of Faecalibacterium prausnitzii in faecal samples from Crohn's disease patients

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years old
* Crohn's disease patients
* Inflammatory activity confirmed by imaging techniques (colonoscopy or magnetic resonance imaging (MRI))
* Refractory inflammatory luminal disease (with or without perianal involvement) at any level of the gastrointestinal tract requiring therapy with adalimumab,according to standard clinical practice.
* Stable maintenance of any other medication (corticosteroids and / or immunosuppressants and/or 5-aminosalicylic acid (5-ASA)) for the past 4 weeks
* Screening tests required for a safe administration of anti tumour necrosis factor (anti-TNF) antibodies will be performed according to standard clinical practice

Exclusion Criteria:

* Subjects consuming prebiotic supplements (inulin, FOS, galactooligosaccharides (GOS)) in their regular diet.
* Antibiotic use within the past 2 months
* Previous anti-TNF therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
FOS increases counts of Faecalibacterium prausnitzii in faecal samples from Crohn's disease patients | 14 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital de Santiago, Santiago de Compostela, A Coruña
  - Hospital de Bellvitge, Hospitalet Del Llobregat, Barcelona
  - Hospital Universitari vall d'Hebron, Barcelona
  - Hospital Josep Trueta, Girona
  - Hospital La Princesa, Madrid